CLINICAL TRIAL: NCT00430261
Title: Phase II Trial of Sunitinib in Bronchoalveolar Carcinoma or Never-Smokers With Any Lung Adenocarcinoma
Brief Title: Phase II Trial of Sunitinib in BAC or Never-Smokers With Any Lung Adenocarcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Swedish Medical Center (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Howard jack West, M.D., Swedish Medical Center, Swedish Cancer Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRC 05160
Record Dates: First submitted 2007-01-30; First posted 2007-02-01 (Estimated); Last update posted 2010-10-06 (Estimated); Status verified 2010-10

CONDITIONS: Lung Cancer; Adenocarcinoma
Keywords: bronchoalveolar carcinoma; BAC; adenocarcinoma; lung cancer; oral; Stage IIIB and IV lung cancer; Any bronchoalveolar carcinoma (BAC); Any adenocarcinoma in a never-smoker
MeSH Terms: conditions — Lung Neoplasms; Adenocarcinoma; Adenocarcinoma, Bronchiolo-Alveolar | interventions — Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: sunitinib — 50mg po qd x 4 weeks on followed by 2 weeks off for a 6 week cycle.
  Other Names: SU011248

SUMMARY:
This is an open-label study of a new oral drug for advanced stage (IIIB or IV) lung cancer. The cancer must be EITHER bronchoalveolar carcinoma (BAC) type, or if the patient is a never-smoker (less than 100 cigarettes lifetime) the cancer can be any type of adenocarcinoma.

DETAILED DESCRIPTION:
To participate in this study, patients must have disease that can be measured on a CT scan. Brain metastases are OK if stable. Pregnant and/or nursing women may not participate. This drug has been approved by the FDA for the treatment of advanced renal cell cancer and a certain type of stomach/intestinal cancer. Its efficacy in lung cancer in currently unknown. Common side effects include fatigue, nausea, diarrhea, skin reaction, and decreased blood counts.

ELIGIBILITY:
Inclusion Criteria:

* Bronchoalveolar carcinoma with disease measurable on CAT scan
* Any lung adenocarcinoma in a never-smoker (less than 100 cigarettes lifetime) with disease measurable on CAT scan
* Stage IIIB or IV

Exclusion Criteria:

* Uncontrolled hypertension
* Unstable brain metastases
* Pregnant/nursing women
* Uncontrolled thyroid disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2007-01; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Progression-Free Survival | January 2009

CONTACTS AND LOCATIONS:
Overall Officials: Howard West, M.D., Principal Investigator — Swedish Cancer Institute
Locations (1):
- Swedish Cancer Institute, Seattle, Washington, United States